CLINICAL TRIAL: NCT03300024
Title: A Prospective Randomized Study of Bovine Carotid Artery Biologic Graft and Expanded Polytetrafluoroethylene for Permanent Hemodialysis Access
Brief Title: Bovine Carotid Artery Biologic Graft and Expanded Polytetrafluoroethylene for Permanent Hemodialysis Access
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00069002
Record Dates: First submitted 2017-09-18; First posted 2017-10-03 (Actual); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: End Stage Renal Disease; Hemolysis; Arteriovenous Graft
Keywords: Hemodialysis; Arteriovenous; Graft; polytetrafluoroethylene; Bovine
MeSH Terms: conditions — Kidney Failure, Chronic; Hemolysis

STUDY DESIGN:
Intervention Model Description: Patients will undergo surgery as per standard of care and receive the randomized graft in compliance to National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines for Arteriovenous graft creation. Surgeries will be elective in nature. The grafts will be placed either in the arm (brachial artery-axillary vein) or forearm (brachial artery to cephalic or suitably sized vein) based on anatomic suitability
Who Masked: Outcomes Assessor
Masking Description: The study will not be blinded because patient side blinding is expected to have minimal to no effect, while physician side blinding is impractical; and difficult to achieve due to the primary surgeon being the one usually who follows up on any intervention or treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Expanded polytetrafluoroethylene (ePTFE) (Active Comparator): The ePTFE grafts used are the Flixene (Maquet-Atrium Medical, Hudson, NH), Advanta VXT (Maquet-Atrium), GORE-TEXStretch Vascular Graft For Vascular Access (W. L. Gore and Associates, Flagstaff, Ariz), or Venaflo (Bard Peripheral Vascular, Tempe, Ariz). The choice of graft used is at the surgeons' discretion. The graft it is offered in both large and small diameters, as well as thin-wall and rapidly-tapering designs for cases where arterial steal syndrome is a potential complication. A 6 mm graft featuring external supporting rings in 5 cm centered or 7 cm offset sections enables tight loop configurations and crossing the cubitus. A 4-7 mm tapered graft with 10 or 15 cm of removable rings allows for tailoring or exact placement of the ringed section.
  Interventions: Device: Expanded polytetrafluoroethylene Graft
- Bovine carotid Artery Graft (Experimental): The bovine carotid artery biological grafts (Artegraft®; Artegraft, Inc., North Brunswick, NJ) consist of a biological fibrous matrix processed to enhance long-term patency and provide a tightly woven, cross-linked conduit that is flexible and compliant.
  Interventions: Device: Bovine Carotid Artery Graft

INTERVENTIONS:
Device: Expanded polytetrafluoroethylene Graft — Group will receive any standard ePTFE graft (control) based on the surgeons' discretion. The graft will be placed either in the arm (brachial artery to axillary vein) or forearm (brachial artery to cephalic or suitably sized vein) depending on which location works best in your particular case.
  Other Names: Synthetic Graft
  Arms: Expanded polytetrafluoroethylene (ePTFE)
Device: Bovine Carotid Artery Graft — Group will receive the BCA graft (experimental).The graft will be placed either in the arm (brachial artery to axillary vein) or forearm (brachial artery to cephalic or suitably sized vein) depending on which location works best in your particular case.
  Other Names: Biological Graft
  Arms: Bovine carotid Artery Graft

SUMMARY:
The investigators propose a randomized study to compare bovine carotid artery (BCA) biologic grafts and expanded polytetrafluoroethylene grafts (ePTFE) for permanent hemodialysis access.

DETAILED DESCRIPTION:
Arteriovenous grafts (AVG) remain reliable substitutes for permanent hemodialysis access in scenarios that preclude the placement of arteriovenous fistulae. There is scarcity of evidence to support the current preference of synthetic conduits over biologic grafts in clinical practice. Advances in the design of AVG's warrant contemporary comparisons between synthetic and biologic AVG options. This is especially important as biologic conduits may confer an advantage by virtue of their inherent similarity to the native human vasculature.

The overall goal of this project is to compare one and two year patency (functional, primary, primary assisted and secondary), complication rates and re-intervention rates between BCA and standard ePTFE grafts. The investigators hypothesize that vascular patient who will receive the BCA graft will have improved patency as well as lower complication and re-intervention rates compared to the standard ePTFE graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Have End Stage Renal Disease and are undergoing Arterio-Venous-Graft surgery
* Not Eligible to receive an Arterio-Venous-Fistula
* Provided written informed consent
* Agreed to return for all required clinical follow up for the study

Exclusion Criteria:

* Eligible to receive an Arterio-Venous-Fistula
* Known allergic reaction or history of intolerance to any ePTFE or BCA components
* Local infection at AVG placement site at the time of surgery
* Patients with a bleeding disorder or who refuse blood transfusion
* Patients with an active malignancy
* Life expectancy less than 1 year
* Pregnant women or those planning on becoming pregnant for the duration of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reifsnyder, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only key study personnel will be responsible for entering and tracking information. At the end of the study period, study coordinators and research fellows will have access to the final trial dataset and will analyse the data. The final results will be communicated to the PI and co-PI's, the sponsors and participants and will be later published in a peer-reviewed scientific journal.

REFERENCES:
- [Derived] Dakour Aridi H, Arhuidese I, Scudder M, Reifsnyder T, Malas MB. A prospective randomized study of bovine carotid artery biologic graft and expanded polytetrafluoroethylene for permanent hemodialysis access. J Vasc Surg. 2018 May;67(5):1606-1612.e4. doi: 10.1016/j.jvs.2017.12.058. Epub 2018 Mar 19. PMID 29567027

RESULTS

PARTICIPANT FLOW:
Groups:
- Expanded Polytetrafluoroethylene (ePTFE): The ePTFE grafts used are the Flixene (Maquet-Atrium Medical, Hudson, NH), Advanta VXT (Maquet-Atrium), GORE-TEXStretch Vascular Graft For Vascular Access (W. L. Gore and Associates, Flagstaff, Ariz), or Venaflo (Bard Peripheral Vascular, Tempe, Ariz). The choice of graft used is at the surgeons' discretion.
  Expanded polytetrafluoroethylene Graft: Group will receive any standard ePTFE graft (control) based on the surgeons' discretion. The graft will be placed either in the arm (brachial artery to axillary vein) or forearm (brachial artery t
- Bovine Carotid Artery Graft: The bovine carotid artery (BCA) biological grafts (Artegraft®; Artegraft, Inc., North Brunswick, NJ) consist of a biological fibrous matrix processed to enhance long-term patency and provide a tightly woven, cross-linked conduit that is flexible and compliant.
  Bovine Carotid Artery Graft: Group will receive the BCA graft (experimental).The graft will be placed either in the arm (brachial artery to axillary vein) or forearm (brachial artery to cephalic or suitably sized vein) depending on which location works best in your particular case.
Period: Overall Study
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Started | 4 | 6
Completed | 0 | 0
Not Completed | 4 | 6
Not completed — Physician Decision | 4 | 6

BASELINE CHARACTERISTICS:
Population: Work on this project was discontinued. Baseline data for "Race and Ethnicity" was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 63.5 [60 to 70] | 67.2 [45 to 80] | 65.7 [45 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Primary Graft Patency
Description: Primary patency is defined as the interval from graft placement to any intervention for stenosis with or without complete occlusion (thrombosis).
Time Frame: One year after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Bovine Carotid Artery Graft | Expanded Polytetrafluoroethylene (ePTFE)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percentage of Patients With Primary-Assisted Graft Patency
Description: Assisted primary patency is defined as the interval from graft placement to the first episode of complete occlusion.
Time Frame: One year after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Percentage of Patients With Secondary Graft Patency
Description: Secondary patency is defined as the interval from graft placement to graft failure.
Time Frame: One year after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Percentage of Patients With Functional Patency
Description: Functional patency represents the interval from the first time the graft is used for hemodialysis to any qualifying event (stenosis, thrombosis, graft failure)
Time Frame: One year after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Percentage of Patients With Primary Graft Patency
Description: as for outcome 1
Time Frame: Two years after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Percentage of Patients With Primary-Assisted Graft Patency
Description: Assisted primary patency is defined as the interval from graft placement to the first episode of complete occlusion.
Time Frame: Two years after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Percentage of Patients With Secondary Graft Patency
Description: Secondary patency is defined as the interval from graft placement to graft failure.
Time Frame: Two years after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Percentage of Patients With Functional Patency
Description: as for outcome 4
Time Frame: Two years after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Incidence of Pseudoaneurysms Formation at the Access Site
Time Frame: At 6 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence of Pseudoaneurysms Formation at the Access Site
Time Frame: At 12 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence of Pseudoaneurysms Formation at the Access Site
Time Frame: At 18 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Incidence of Pseudoaneurysms Formation at the Access Site
Time Frame: At 24 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Patients With Surgical Site Infection
Description: The presence of erythema or purulent drainage at the surgical incision and need for intravenous antibiotics or surgical intervention.
Time Frame: At 6 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Patients With Surgical Site Infection
Description: as for outcome 13
Time Frame: At 12 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Patients With Surgical Site Infection
Description: as for outcome 13
Time Frame: At 18 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage of Patients With Surgical Site Infection
Description: as for outcome 13
Time Frame: At 24 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Steal Syndrome
Description: Steal syndrome will be staged per standard as follows: Stage I: pale/blue and/or cold hand without pain; Stage II: Pain during exercise and/or hemodialysis; Stage III: Rest pain; Stage IV: Ulcers/necrosis/gangrene. Accordingly, surgical intervention will be carried out for patients with stage III or IV steal.
Time Frame: At 6 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Steal Syndrome
Description: as for outcome 17
Time Frame: At 12 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Steal Syndrome
Description: as for outcome 17
Time Frame: At 18 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Steal Syndrome
Description: as for outcome 17
Time Frame: At 24 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Percentage of Patients Requiring Revisional Procedures of the Arteriovenous Graft
Description: At hemodialysis, the grafts will be accessed with 15 or 17 gauge needles inserted at any angle between 25-30 degrees (the same method used for a native arterio-venous fistula). If by physical examination the graft is thrombosed, then the patient will immediately be referred for endovascular thrombectomy and revision. If the graft is patent, but problematic, the patient will be referred for an urgent fistulogram and endovascular reintervention
Time Frame: At 6 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Percentage of Patients Requiring Revisional Procedures of the Arteriovenous Graft
Description: as for outcome 21
Time Frame: At 12 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percentage of Patients Requiring Revisional Procedures of the Arteriovenous Graft
Description: as for outcome 21
Time Frame: At 18 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Percentage of Patients Requiring Revisional Procedures of the Arteriovenous Graft
Description: as for outcome 21
Time Frame: At 24 months after Graft Placement
Population: Data was not collected for this outcome measure
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable. Work on this project was discontinued. No adverse event data was collected.
Description: No adverse event data was collected.
Arm/Group | Expanded Polytetrafluoroethylene (ePTFE) | Bovine Carotid Artery Graft
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03300024/Prot_SAP_002.pdf
  • Informed Consent Form (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03300024/ICF_003.pdf